CLINICAL TRIAL: NCT03164109
Title: A Phase 1, Randomized, Placebo-and Positive-Controlled Crossover Study to Determine the Effect of Single-Dose GC4419 on QTc Interval in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galera Therapeutics, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GTI-4419-002
Record Dates: First submitted 2017-05-15; First posted 2017-05-23 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers; Healthy
Keywords: Healthy Adult; Superoxide Dismutase; Free Radical Dismutase; Cardiodynamic Assessment
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- GC4419 IV (Experimental)
  Interventions: Drug: GC4419 IV
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Oral moxifloxacin (Active Comparator)
  Interventions: Drug: Oral moxifloxacin

INTERVENTIONS:
Drug: GC4419 IV — 50mg infused IV over 15 minutes
  Arms: GC4419 IV
Drug: Placebo — Infused IV over 15 minutes
  Arms: Placebo
Drug: Oral moxifloxacin — 400 mg tablet orally with 250 mL room temperature water
  Arms: Oral moxifloxacin

SUMMARY:
This is a partially double-blind study in healthy adult subjects, which will be conducted as a placebo- and active-controlled, single-dose, crossover study.

Twenty-eight subjects will be enrolled to ensure 24 subjects on all study periods. All subjects will receive all 3 study treatments (GC4419, placebo and moxifloxacin) in randomized sequence.

Cardiodynamic assessment using continuous ECG recordings (Holters) will be performed for approximately 26 hours on the day of dosing (Day 1) in each study period. ECGs will be extracted serially pre- and post-dose and predefined timepoints at which subjects will be supinely resting.

Subjects will be supinely resting for at least 10 minutes prior to and 5 minutes after each nominal timepoint for ECG extraction.

Blood draws for PK will be performed in all periods at the same timepoints and always after ECG extraction.

Subjects will be domiciled in the clinic from noon/afternoon of the day before dosing (Day -1) until completion of safety procedures on Day 2 in each study period.

All subjects (including subjects who terminate the study early) will return to the clinical research unit (CRU) 14 (± 1) days after the last administration of study treatment for follow-up procedures and to determine if any Adverse Event (AE) has occurred since the last study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female, 18-55 years of age
2. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dose.
3. Must weigh at least 60 kg for males or 52 kg for females and have a body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or ECGs
5. For a female of childbearing potential: either be sexually inactive as a voluntary lifestyle choice for at least 1 year prior to first dosing until 21 days following last dosing or be using an acceptable birth control method
6. For a female of non-childbearing potential: must have undergone an acceptable sterilization procedure or be postmenopausal for at least 1 year prior to the first dose
7. Willing and able to comply with the protocol.
8. Seated blood pressure between 90/40 mmHg and 140/90 mmHg
9. Has serum potassium, calcium, and magnesium levels within the normal range at screening.

Exclusion Criteria:

1. History or presence of clinically significant medical or psychiatric condition, disease or illness
2. History or presence of alcoholism or drug abuse within the past 2 years
3. History or presence of hypersensitivity to the study drugs
4. History of significant multiple and/or severe allergies
5. Female subjects who are pregnant or lactating.
6. Positive results at screening for human immunodeficiency virus (HIV), syphilis, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
7. Unable to refrain from or anticipates the use of any drug, including prescription and non-prescription medications 14 days prior to the first dose of study drug and throughout the study.
8. Any drugs known to be significant inhibitors or inducers of CYP enzymes and/or P-gp, including St. John's Wort, for 28 days prior to the first dose of study drug and throughout the study.
9. Has been on a diet incompatible with the on-study diet, within the 28 days prior to the first dose of study drug, and throughout the study.
10. Donation of blood or significant blood loss within 56 days
11. Plasma donation within 7 days prior to the first dose of study drug.
12. Has had surgery or any medical condition which may affect the absorption, distribution, metabolism, or elimination of the study drug within 6 months.
13. Participation in another clinical trial within 28 days
14. Participation in a previous clinical trial where subject received GC4419.
15. History or presence of: hypokalemia, risk factors for Torsades de Pointes , sick sinus syndrome, second, or third degree atrioventricular block, myocardial infarction, pulmonary congestion, cardiac arrhythmia, prolonged QT interval, or conduction abnormalities; repeated or frequent syncope or vasovagal episodes; hypertension, angina, bradycardia, or severe peripheral arterial circulatory disorders.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

PRIMARY OUTCOMES:
Change in QT interval corrected for heart rate using the Fridericia formula (QTcF) | From 45 minute pre-dose to 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Jon T Holmlund, MD, Study Chair — Galera Therapeutics
Locations (1):
- Nucleus Network Limited, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No